CLINICAL TRIAL: NCT06761976
Title: An Expanded Access Program to Provide Oral Sevabertinib (BAY 2927088) in Adult Participants With Locally Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC) Harboring an HER2 (Human Epidermal Growth Factor Receptor 2) Activating Mutation
Brief Title: Expanded Access to Provide Sevabertinib (BAY 2927088) for the Treatment of Locally Advanced or Metastatic NSCLC With HER2 Mutation
Status: Available | Type: Expanded Access
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 22913; 22978 (Other: Bayer ID)
Record Dates: First submitted 2024-12-30; First posted 2025-01-07 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Advanced Non-small Cell Lung Cancer; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: Sevabertinib — Sevabertinib is self-administered by the patient BID (twice a day) as tablets for oral administration
  Other Names: BAY2927088

SUMMARY:
The purpose of this Expanded Access Program (EAP) is to provide access to sevabertinib, for participants previously treated with locally advanced or metastatic non-small cell lung cancer (NSCLC) with mutations in the human epidermal growth factor receptor 2 (HER2) gene, which have no other therapeutic option.

ELIGIBILITY:
Inclusion Criteria

* Signed and dated written informed consent
* Age ≥18 years
* Histologically or cytologically confirmed locally advanced or metastatic NSCLC
* Documented disease progression after treatment with at least one prior systemic therapy for advanced disease
* Documented HER2 activating mutation
* Expected minimum life expectancy of 12 weeks
* Performance status of 0 or 1
* Participants must be able to take oral medication
* Blood test results within certain ranges
* Adequate coagulation as assessed by lab tests or on stable anticoagulation treatment
* Adequate cardiac function
* Negative serum pregnancy test in women of childbearing potential within 72 hours of the first dose
* Ability to receive prescription of loperamide from the treating physician

Exclusion Criteria

* Investigational agent or anticancer therapy within 2 weeks prior to planned start of sevabertinib or 5 half-lives, whichever is shorter, and without recovery of clinically significant toxicities from that therapy
* Prior progression while receiving approved or investigational tyrosine kinase inhibitors targeting HER2
* Symptomatic or unstable brain metastases
* Treatment with immunotherapy ≤ 28 days prior to the first dose of IMP
* Past medical history of Grade ≥2 ILD, drug-induced interstitial lung disease
* Inability to discontinue treatment with a strong CYP3A4 inhibitor or inducer prior to start of treatment initiation
* Any uncontrolled intercurrent illness or condition including, but not limited to, uncompensated respiratory, cardiac, hepatic, or renal disease, ongoing or active infection (including active clinical tuberculosis), renal transplant or psychiatric illness/social situations that would limit compliance
* Pregnancy or lactation
* History of clinically significant cardiac disease

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

REFERENCES:
- See also: Click here for access to information about the study and about Bayer's transparency standards. — https://clinicaltrials.bayer.com/study/22913